CLINICAL TRIAL: NCT04680637
Title: A Phase 2b Dose Ranging Study to Evaluate the Efficacy and Safety of Efavaleukin Alfa in Subjects With Active Systemic Lupus Erythematosus With Inadequate Response to Standard of Care Therapy
Brief Title: Efficacy and Safety of Efavaleukin Alfa in Subjects With Active Systemic Lupus Erythematosus
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The trial was terminated prematurely as it met pre-defined criteria for futility at IA3.
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20200234
Record Dates: First submitted 2020-12-18; First posted 2020-12-23 (Actual); Results first posted 2024-06-28 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Active Systemic Lupus Erythematosus
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo + Standard of Care (Placebo Comparator)
  Interventions: Drug: Placebo; Other: Standard of Care
- Efavaleukin Alfa Dose Level One + Standard of Care (Experimental)
  Interventions: Drug: Efavaleukin Alfa; Other: Standard of Care
- Efavaleukin Alfa Dose Level Two + Standard of Care (Experimental)
  Interventions: Drug: Efavaleukin Alfa; Other: Standard of Care
- Efavaleukin Alfa Dose Level Three + Standard of Care (Experimental)
  Interventions: Drug: Efavaleukin Alfa; Other: Standard of Care

INTERVENTIONS:
Drug: Efavaleukin Alfa — Administered as a subcutaneous (SC) injection.
  Other Names: AMG 592
  Arms: Efavaleukin Alfa Dose Level One + Standard of Care; Efavaleukin Alfa Dose Level Three + Standard of Care; Efavaleukin Alfa Dose Level Two + Standard of Care
Drug: Placebo — Administered as a subcutaneous (SC) injection.
  Arms: Placebo + Standard of Care
Other: Standard of Care — Standard of care procedures and therapies for managing active systemic lupus erythematosus will be carried out according to each investigator's standard procedures.

SUMMARY:
The primary objective is to evaluate the efficacy and safety of efavaleukin alfa in subjects with active systemic lupus erythematosus.

ELIGIBILITY:
Inclusion Criteria:

* Participant has provided informed consent prior to initiation of any study specific activities/procedures.
* Participant is aged between 18 and 75.
* Fulfills classification criteria for systemic lupus erythematosus (SLE) according to the 2019 European League Against Rheumatism (EULAR)/American College of Rheumatology (ACR) classification criteria for SLE with antinuclear antibody ≥ 1:80 by immunofluorescence on Hep-2 cells being present at screening.
* Hybrid SLEDAI score ≥ 6 points with a "Clinical" hSLEDAI score ≥ 4 points. The "Clinical" hSLEDAI is the hSLEDAI assessment score without the inclusion of points attributable to laboratory results, including urine or immunologic parameters.
* British-Isles Lupus Assessment Group (BILAG) index score (BILAG 2004) of ≥ 1 A item or ≥ 2 B items.
* Must be taking ≥ 1 of the following SLE treatments (or regional equivalent): hydroxychloroquine, chloroquine, quinacrine, mycophenolate mofetil, azathioprine, methotrexate, dapsone, or oral calcineurin inhibitors, or OCS. A participant may enter the study on OCS alone (prednisone ≥ 10 mg/day or equivalent) only if the participant has previously documented trial of anti-malarial or immunosuppressant treatment for SLE. Participants must be on a stable dose for ≥ 8 weeks prior to screening for all antimalarials and immunosuppressants, with the exception of OCS doses which must be stable for ≥ 2 weeks prior to screening.
* For participants taking OCS, dose must be ≤ 20 mg/day of prednisone or OCS equivalent, and the dose must be stable at baseline visit and for ≥ 2 weeks prior to screening visit.
* Stability of SLE treatments: OCS and other immunosuppressants/immunomodulator agents and doses must be stable since screening visit.
* Disease activity: active disease as indicated by clinical hSLEDAI score ≥ 4 must be observed (clinical hSLEDAI score is the hSLEDAI assessment score without the inclusion of points attributable to laboratory results including urine and immunologic parameters).

Exclusion Criteria:

* Lupus nephritis if any of the following are present: urine protein creatinine ratio ≥ 2000 mg/g (or equivalent) at screening, OR requiring induction therapy currently or within 1 year prior to screening, OR histological evidence (if available) of diffuse proliferative glomerulonephritis within 12 weeks prior to screening.
* Active CNS lupus within 1 year prior to screening including, but not limited to, aseptic meningitis, ataxia, CNS vasculitis, cranial neuropathy, demyelinating syndrome, optic neuritis, psychosis, seizures, or transverse myelitis.
* Currently present or within 1 year prior to screening a diagnosis of any chronic inflammatory disease other than SLE (eg, rheumatoid arthritis) which would interfere with SLE disease assessment.
* History of any disease other than SLE that has required treatment with oral or parenteral corticosteroids for > 2 weeks within 4 months prior to screening.
* Active infection (including chronic or localized infections) for which anti-infectives are indicated currently or within 4 weeks prior to screening visit OR presence of serious infection, defined as requiring hospitalization or intravenous anti-infectives within 8 weeks prior to screening visit.
* Active tuberculosis or latent tuberculosis with no documented past history of adequate treatment per local standard of care.
* Positive test for tuberculosis during creening defined as: either a positive or indeterminate QuantiFERON®-TB or T-spot test OR positive purified protein derivative (PPD) (≥5 mm of induration at 48 to 72 hours after test is placed).
* Positive for hepatitis B surface antigen (HBsAg); or positive for hepatitis B core antibody (HBcAb). A history of hepatitis B vaccination without history of hepatitis B infection (ie, positive hepatitis B surface antibody (HBsAb), negative HBsAg and negative HBcAb) is allowed.
* Positive for hepatitis C antibody.
* Known history of HIV or positive HIV test at screening.
* Presence of 1 or more significant concurrent medical conditions, including but not limited to the following:

  * poorly controlled diabetes (hemoglobin A1C > 7) or hypertension
  * symptomatic heart failure (New York Heart Association class III or IV)
  * myocardial infarction or unstable angina pectoris within the past 12 months prior to screening
  * severe chronic pulmonary disease requiring oxygen therapy
  * multiple sclerosis or any other demyelinating disease
* Any history of malignancy with the following exceptions:
* resolved non-melanoma skin cancers > 5 years prior to screening
* resolved cervical carcinoma > 5 years prior to screening
* resolved breast ductal carcinoma in situ > 5 years of screening
* Currently receiving or had treatment with: cyclophosphamide, chlorambucil, nitrogen mustard, or any other alkylating agent within 6 months prior to screening or sirolimus within 4 weeks prior screening.
* Currently receiving or had treatment with a Janus kinase (JAK) inhibitor within 3 months or less than 5 drug half-lives (whichever is longer) prior to screening.
* Currently receiving or had treatment with an immune checkpoint inhibitor (eg, programmed death 1 [PD-1] inhibitor, programmed death ligand 1 [PD-L1] inhibitor, cytotoxic T-lymphocyte associated protein 4 [CTLA-4] inhibitor).

Note: Abatacept is not considered a CTLA-4 inhibitor and is referred to below.

* Currently receiving or had treatment within 12 months prior to screening with T-cell depleting agents (eg, antithymocyte globulin, Campath).
* Currently receiving of had treatment with an interleukin 2 (IL-2) based therapy (eg, Proleukin).
* Current or previous treatment with a biologic agent with immunosuppressive/immunomodulatory activity as follows: rituximab within 6 months prior to screening; abatacept and belimumab within the past 3 months prior to screening; other biologics within < 5 drug half lives prior to screening.
* Participants who have received intraarticular, intralesional, or intramuscular corticosteroids within 2 weeks prior to screening or intravenous corticosteroids within 6 weeks prior to screening.
* Participants who have received live vaccines within 5 weeks prior to screening, or plan to receive live vaccines during the treatment period and up to 6 weeks after the end of treatment period in the study.
* Currently receiving treatment in another investigational device or drug study.
* Ending a treatment with an investigational drug or investigational device less than 3 months or 5 half-lives from the last dose of the investigational drug (whichever is longer) at screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2021-05-06 (Actual); Primary Completion 2023-05-22 (Actual); Study Completion 2023-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (150):
- United States (51):
  - University of Alabama at Birmingham,Arthritis Clinical Intervention Program, Birmingham, Alabama
  - Arizona Arthritis and Rheumatology Associates PC, Gilbert, Arizona
  - Arizona Arthritis And Rheumatology Associates PC, Glendale, Arizona
  - Arizona Arthritis and Rheumatology Associates PC, Tucson, Arizona
  - Loma Linda University Health Care, Loma Linda, California
  - University of California Los Angeles, Los Angeles, California
  - University of California Irvine, Orange, California
  - Robin K Dore MD Inc, Tustin, California
  - Arthritis and Rheumatic Disease Specialties, Aventura, Florida
  - Life Clinical Trials, Aventura, Florida
  - Centre for Rheumatology Immunology and Arthritis, Fort Lauderdale, Florida
  - GNP Research, Hollywood, Florida
  - Millennium Research, Ormond Beach, Florida
  - Integral Rheumatology and Immunology Specialists, Plantation, Florida
  - Suncoast Medical Clinic, St. Petersburg, Florida
  - Baycare Medical Group Inc, Tampa, Florida
  - University of Chicago, Chicago, Illinois
  - Greater Chicago Specialty Physicians, Schaumburg, Illinois
  - Clinic of Robert Hozman, MD - Clinical Investigational Specialists, Inc, Skokie, Illinois
  - Western Kentucky Rheumatology PLLC, Hopkinsville, Kentucky
  - Accurate Clinical Research, Lake Charles, Louisiana
  - Michigan Rheumatology Group, PC - Grand Blanc Office, Grand Blanc, Michigan
  - Arthritis and Rheumatology of Michigan, Lansing, Michigan
  - New York University Langone Ambulatory Care Brooklyn Heights, Brooklyn, New York
  - Feinstein Institute for Medical Research, Manhasset, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Institute for Clinical and Translation Research at Einstein and Montefiore Clinical Research Center, The Bronx, New York
  - University of North Carolina at Chapel Hill Thurston Arthritis Research Center, Chapel Hill, North Carolina
  - Joint and Muscle Research Institute, Charlotte, North Carolina
  - DJL Clinical Research PLLC, Charlotte, North Carolina
  - Javara, Charlotte, North Carolina
  - Atrium Health Rheumatology, Charlotte, North Carolina
  - Arthritis and Rheumatology Center of Oklahoma PLLC, Oklahoma City, Oklahoma
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - University of Pittsburgh Medical Center Lupus Center of Excellence, Pittsburgh, Pennsylvania
  - Columbia Arthritis Center, PA, Columbia, South Carolina
  - Piedmont Arthritis Clinic, Greenville, South Carolina
  - West Tennessee Research Institute, LLC, Jackson, Tennessee
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Ramesh C Gupta MD, Memphis, Tennessee
  - Arthritis and Rheumatology Institute, Allen, Texas
  - Precision Comprehensive Clinical Research Solutions, Colleyville, Texas
  - Texas Arthritis Center PA, El Paso, Texas
  - Biopharma Informatic, LLC, Houston, Texas
  - Accurate Clinical Management, Houston, Texas
  - Laila A Hassan, MD, PA, Houston, Texas
  - Trinity Universal Research Associates, LLC, Plano, Texas
  - Clinical Trials of Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio Medical Arts Research Clinic Marc, San Antonio, Texas
  - Arthritis and Osteoporosis Clinic, Waco, Texas
- Medizinische Universitaet Graz, Graz, Austria
- Bulgaria (4):
  - Diagnostic-Consultative Center Sveti Georgi EOOD, Plovdiv
  - Medical Center Excelsior OOD, Sofia
  - Medical Center Academy EOOD, Sofia
  - University Multiprofile Hospital for Active Treatment Sveti Ivan Rilski EAD, Sofia
- Toronto Western Hospital, Toronto, Ontario, Canada
- Chile (8):
  - Investigacion y Terapias Reumatologicas Innovadoras LTDA - Interin LTDA, Providencia, Santiago Metropolitan
  - Enroll SpA, Providencia, Santiago Metropolitan
  - Sociedad de prestaciones Medicas y Paramedicas Goecke Gatica y Compania Limitada - Prosalud, Providencia, Santiago Metropolitan
  - Corporacion de Beneficiencia Osorno, Osorno
  - Estudios Clinicos Limitada - Centro de Estudios Reumatologicos, Santiago
  - CECIM, Santiago
  - Sociedad de Prestaciones Medicas Intermedica Limitada, Valdivia
  - Oncocentro Apys, Viña del Mar
- Colombia (6):
  - Hospital Pablo Tobon Uribe, Medellín, Antioquia
  - Centro Integral de Reumatología del Caribe Circaribe SAS, Barranquilla, Atlántico
  - Centro de Investigacion en Reumatologia y Especialidades Medicas SAS, Bogota, Cundinamarca
  - Solano y Terront Servicios Medicos Ltda - Uniendo, Bogota, Cundinamarca
  - Mediservis del Tolima IPS SAS, Ibagué, Tolima Department
  - Centro Medico Julian Coronel, Cali, Valle del Cauca Department
- France (4):
  - Centre Hospitalier Universitaire de Montpellier Hopital Lapeyronie, Montpellier
  - Centre Hospitalier Universitaire de Strasbourg - Nouvel Hopital Civil, Strasbourg
  - Centre Hospitalier Universitaire de Toulouse - Hopital Rangueil, Toulouse
  - Centre Hospitalier Universitaire de Nancy - Hopital de Brabois, Vandœuvre-lès-Nancy
- Greece (7):
  - Athens Naval Hospital, Athens
  - Laiko General Hospital, Athens
  - Attiko Hospital, Athens
  - University Hospital of Heraklion, Heraklion
  - Olympion Hospital-General Clinic of Patras AE, Pátrai
  - Euromedica - Kyanous Stavros, Thessaloniki
  - Ippokrateio Hospital of Thessaloniki, Thessaloniki
- Tuen Mun Hospital, New Territories, Hong Kong
- Italy (8):
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Università degli studi della Campania Luigi Vanvitelli, Napoli
  - Azienda Ospedaliera di Padova, Padua
  - Azienda Ospedaliera Policlinico Umberto I, Roma
  - Policlinico Universitario Agostino Gemelli, Roma
  - Azienda Ospedaliera Ordine Mauriziano di Torino, Torino
  - Azienda Ospedaliero Universitaria Integrata Santa Maria della Misericordia, Udine
  - Centro Ricerche Cliniche, Verona
- Japan (19):
  - Japan Community Healthcare Organization Chukyo Hospital, Nagoya, Aichi-ken
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - National Hospital Organization Chibahigashi National Hospital, Chiba, Chiba
  - Hospital of the University of Occupational and Environmental Health Japan, Kitakyushu-shi, Fukuoka
  - Hiroshima University Hospital, Hiroshima, Hiroshima
  - Sapporo City General Hospital, Sapporo, Hokkaido
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Eiraku Clinic, Kagoshima, Kagoshima-ken
  - Kagoshima University Hospital, Kagoshima, Kagoshima-ken
  - St Marianna University Hospital, Kawasaki-shi, Kanagawa
  - National University Corporation Tohoku University Tohoku University Hospital, Sendai, Miyagi
  - Nagasaki University Hospital, Nagasaki, Nagasaki
  - Seirei Hamamatsu General Hospital, Hamamatsu, Shizuoka
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - St Lukes International Hospital, Chuo-ku, Tokyo
  - National Hospital Organization Tokyo Medical Center, Meguro-ku, Tokyo
  - Keio University Hospital, Shinjuku-ku, Tokyo
  - Center Hospital of the National Center for Global Health and Medicine, Shinjuku-ku, Tokyo
- Mexico (6):
  - Centro Integral en Reumatologia SA de CV, Guadalajara, Jalisco
  - Centro de Estudios de Investigacion Basica y Clinica, Sc, Guadalajara, Jalisco
  - CITER SA de CV (Centro de Investigación y Tratamiento de las Enfermedades Reumáticas SA de CV), Mexico City, Mexico City
  - Eukarya Pharmasite sc, Monterrey, Nuevo León
  - Centro de Investigacion Integral Medivest SC, Chihuahua City
  - Phylasis Clínicas Research S. De R. L. De C. V., Cuautitlán Izcalli
- Poland (6):
  - Centrum medyczne intercore sp zoo, Bydgoszcz
  - Centrum Medyczne Pratia Czestochowa, Częstochowa
  - Centrum Badan Klinicznych Wojciech Brzezicki, Malbork
  - NZOZ Lecznica MAK-MED sc, Nadarzyn
  - Gabinety Lekarskie RIVERMED, Poznan
  - Reumatop Grzegorz Rozumek, Karin Pistorius, Wroclaw
- Russia (6):
  - Limited liability company Scientific Research Medical Complex Your Health, Kazan'
  - FSBSI SRI of Rheumatology na V A Nasonova, Moscow
  - I M Sechenov First Medical University of the MoH of RF, Moscow
  - Saint-Petersburg State Budget Healthcare Institution Clinical Rheumatology Hospital 25, Saint Petersburg
  - LLC Medical Sanitary Unit №157, Saint Petersburg
  - Center for medical consultations and research - practice, Yaroslavl
- South Korea (4):
  - Daegu Catholic Universtiy Medcial Center, Daegu
  - Seoul National University Hospital, Seoul
  - Hanyang University Seoul Hospital, Seoul
  - Ajou University Hospital, Suwon-si, Gyeonggi-do
- Spain (8):
  - Hospital Universitario Reina Sofia, Córdoba, Andalusia
  - Hospital Infanta Luisa, Seville, Andalusia
  - Hospital Universitario Araba, Vitoria-Gasteiz, Basque Country
  - Hospital Universitario Hospiten Rambla, Santa Cruz de Tenerife, Canary Islands
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia
  - Corporacio Sanitaria Parc Tauli, Sabadell, Catalonia
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela, Galicia
  - Hospital Universitari i Politecnic La Fe, Valencia, Valencia
- Switzerland (2):
  - Universitaetsspital Basel, Basel
  - Kantonsspital St Gallen, Sankt Gallen
- Taiwan (4):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Chung Shan Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
- Turkey (Türkiye) (4):
  - Cukurova Universitesi Balcali Hastanesi Saglik Uygulama ve Arastirma Merkezi, Adana
  - Hacettepe Universitesi Tip Fakultesi, Ankara
  - Akdeniz Universitesi Tip Fakultesi, Antalya
  - Istanbul Universitesi Istanbul Tip Fakultesi, Istanbul

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Derived] Garces S, Karis E, Merrill JT, Askanase AD, Kalunian K, Mo M, Milmont CE. Improving resource utilisation in SLE drug development through innovative trial design. Lupus Sci Med. 2023 Jul;10(2):e000890. doi: 10.1136/lupus-2022-000890. PMID 37491104
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 73 centers in 13 countries (Bulgaria, Chile, Colombia, Greece, Italy, Japan, Mexico, Poland, Russian Federation, Spain, Switzerland, Taiwan, and the United States) between 06 May 2021 and 24 May 2023.
Pre-assignment Details: A total of 464 participants were screened, of which 168 participants were enrolled and received efavaleukin alfa.
Groups:
- Placebo: Participants received placebo matching efavaleukin alfa every two weeks (Q2W) through a subcutaneous (SC) injection for up to 52 weeks.
- Efavaleukin Alfa Low Dose: Participants received low dose efavaleukin alfa Q2W through a SC injection for up to 52 weeks.
- Efavaleukin Alfa Medium Dose: Participants received medium dose efavaleukin alfa Q2W through a SC injection for up to 52 weeks.
- Efavaleukin Alfa High Dose: Participants received high dose efavaleukin alfa Q2W through a SC injection for up to 52 weeks.
Period: Overall Study
Arm/Group | Placebo | Efavaleukin Alfa Low Dose | Efavaleukin Alfa Medium Dose | Efavaleukin Alfa High Dose
Started | 41 | 35 | 34 | 58
Received Study Treatment | 41 | 35 | 34 | 58
Completed | 12 | 9 | 10 | 10
Not Completed | 29 | 26 | 24 | 48
Not completed — Lost to Follow-up | 0 | 1 | 0 | 1
Not completed — Death | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 7 | 10 | 17 | 15
Not completed — Decision by Sponsor | 21 | 15 | 7 | 32

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: Included all participants randomized in the study.
Groups:
- Placebo: Participants received placebo matching efavaleukin alfa Q2W through a SC injection for up to 52 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | Efavaleukin Alfa Low Dose | Efavaleukin Alfa Medium Dose | Efavaleukin Alfa High Dose | Total
Number analyzed (Participants) | 41 | 35 | 34 | 58 | 168
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.1 (10.3) | 46.1 (12.8) | 40.3 (12.2) | 42.3 (11.2) | 44.1 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 31 | 33 | 56 | 158
  Male | 3 | 4 | 1 | 2 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 11 | 12 | 22 | 59
  Not Hispanic or Latino | 27 | 24 | 22 | 36 | 109
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 2 | 3 | 5 | 14
  Asian | 6 | 2 | 5 | 6 | 19
  Black (or African American) | 5 | 8 | 1 | 9 | 23
  Multiple | 0 | 0 | 1 | 0 | 1
  White | 25 | 20 | 20 | 29 | 94
  Other | 1 | 3 | 4 | 9 | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieved a Systemic Lupus Erythematosus Responder Index 4 (SRI-4) Response at Week 52
Description: A participant achieved an SRI-4 response if all the following criteria were met:
  * ≥ 4-point reduction from baseline in Hybrid Systemic Lupus Erythematosus Disease Activity Index (hSLEDAI) score (scale 0-105, with higher scores indicating more disease activity).
  * No new British-Isles Lupus Assessment Group (BILAG) A score and no > 1 new BILAG B organ domain scores compared with baseline. The BILAG index evaluates disease activity in 9 separate organ systems. Each of the organ systems are allocated an alphabetical score of A (most active), B (moderate activity), C (minor activity), D (stable) or E (never present).
  * < 0.3-points deterioration from baseline in Physician Global Assessment (PGA) visual analogue (VAS) score (scale 0 to 3, with higher scores indicating more severe disease).
  Participants were considered non-responders for using more than protocol-permitted therapies.
Time Frame: Week 52
Population: Full Analysis Set: Included all participants randomized in the study. Only participants who had the opportunity to complete the visit by the date of the study termination decision being communicated to sites were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Efavaleukin Alfa Low Dose | Efavaleukin Alfa Medium Dose | Efavaleukin Alfa High Dose
Number analyzed (Participants) | 15 | 16 | 17 | 14
Participants | 8 | 4 | 6 | 5

2. Secondary Outcome: Number of Participants Who Achieved a BILAG-based Composite Lupus Assessment (BICLA) Response at Week 52
Description: A participant achieved a BICLA response if all the following criteria were met:
  * At least 1 gradation of improvement in baseline BILAG domain scores in all body systems with moderate or severe disease activity at entry and no > 1 BILAG B domain scores compared with baseline. The BILAG index evaluates disease activity in 9 separate organ systems. Each of the organ systems are allocated an alphabetical score of A (most active), B (moderate activity), C (minor activity), D (stable) or E (never present).
  * No worsening of the hSLEDAI score from baseline (scale 0-105, with higher scores indicating more disease activity).
  * < 0.3-points deterioration from baseline in PGA VAS (scale 0 to 3, with higher scores indicating more severe disease).
  * No initiation of non-protocol treatment.
Time Frame: Week 52
Population: Full Analysis Set: Included all participants randomized in the study. Only participants who had the opportunity to complete the visit by the date of the study termination decision being communicated to sites were included. Participants were considered non-responders for using more than protocol-permitted therapies.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Efavaleukin Alfa Low Dose | Efavaleukin Alfa Medium Dose | Efavaleukin Alfa High Dose
Number analyzed (Participants) | 15 | 16 | 17 | 14
Participants | 6 | 2 | 4 | 4

3. Secondary Outcome: Number of Participants Who Achieved a Lupus Low Disease Activity State (LLDAS) Response at Week 52
Description: A participant achieved an LLDAS response if all the following criteria were met:
  * hSLEDAI ≤ 4 (scale 0-105, higher scores indicating more disease activity) with no activity in major organ systems (renal [proteinuria, hematuria, pyuria, urinary casts], central nervous system [seizure, psychosis, organic brain syndrome, cranial nerve disorder, cerebrovascular accident], cardiopulmonary [pericarditis, pleurisy], vasculitis and fever) & no hemolytic anemia or gastrointestinal activity in BILAG. The BILAG index evaluates disease activity in 9 separate organ systems. Each of the organ systems are allocated an alphabetical score of A (most active) to E (never present).
  * No new lupus disease activity compared with previous assessment defined as no new descriptor scores in hSLEDAI.
  * A score of < 1 in PGA VAS score (scale 0 to 3, with higher scores indicating more severe disease).
  * Current prednisolone dose ≤ 7.5 mg daily.
  * No increase or initiation of immunosuppressive drugs.
Time Frame: Week 52
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Efavaleukin Alfa Low Dose | Efavaleukin Alfa Medium Dose | Efavaleukin Alfa High Dose
Number analyzed (Participants) | 15 | 16 | 17 | 14
Participants | 2 | 3 | 3 | 1

4. Secondary Outcome: Number of Participants With a Reduction of Oral Corticosteroids (OCS) to ≤ 7.5 mg/Day by Week 44 and Sustained Through Week 52 in Participants With a Baseline OCS Dose ≥ 10 mg/Day
Description: Participants taking OCS could begin tapering OCS after the Week 12 assessment up to the Week 44 assessment with initiation of tapering based upon clinical judgement of the treating physician. The tapering schedule was at the discretion of the investigator but should not have been tapered more than 20% of the prior dose per week. Tapering OCS before Week 12 was not encouraged but may have been allowed based upon investigator's judgement. Between weeks 44 and 52, the OCS dosing must again have remained stable.
Time Frame: Baseline to Week 52
Population: Full Analysis Set: Included all participants randomized in the study. Only participants with a baseline OCS dose ≥ 10 mg/day and had the opportunity to complete the visit by the date of the study termination decision being communicated to sites were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Efavaleukin Alfa Low Dose | Efavaleukin Alfa Medium Dose | Efavaleukin Alfa High Dose
Number analyzed (Participants) | 9 | 9 | 8 | 7
Participants | 0 | 1 | 2 | 0

5. Secondary Outcome: Number of Participants Who Achieved a SRI-4 Response at Week 24
Description: A participant achieved an SRI-4 response if all the following criteria were met:
  * ≥ 4-point reduction from baseline in hSLEDAI score (scale 0-105, with higher scores indicating more disease activity).
  * No new BILAG A score and no > 1 new BILAG B organ domain scores compared with baseline. The BILAG index evaluates disease activity in 9 separate organ systems. Each of the organ systems are allocated an alphabetical score of A (most active), B (moderate activity), C (minor activity), D (stable) or E (never present).
  * < 0.3-points deterioration from baseline in PGA VAS score (scale 0 to 3, with higher scores indicating more severe disease).
  Participants were considered non-responders for using more than protocol-permitted therapies.
Time Frame: Week 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Efavaleukin Alfa Low Dose | Efavaleukin Alfa Medium Dose | Efavaleukin Alfa High Dose
Number analyzed (Participants) | 34 | 29 | 31 | 44
Participants | 20 | 13 | 13 | 21

6. Secondary Outcome: Number of Participants Who Achieved a BICLA Response at Week 24
Description: as for outcome 2
Time Frame: Week 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Efavaleukin Alfa Low Dose | Efavaleukin Alfa Medium Dose | Efavaleukin Alfa High Dose
Number analyzed (Participants) | 34 | 29 | 31 | 44
Participants | 17 | 12 | 5 | 17

7. Secondary Outcome: Number of Participants With a hSLEDAI Response at Week 24 and Week 52
Description: The hSLEDAI is a global index that evaluates disease activity and includes both laboratory and clinical parameters. The score ranges from 0 to 105, with higher scores indicating more disease activity.
  A participant achieved a hSLEDAI response if there was a ≥ 4-point reduction in hSLEDAI from baseline.
Time Frame: Week 24 and Week 52
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Efavaleukin Alfa Low Dose | Efavaleukin Alfa Medium Dose | Efavaleukin Alfa High Dose
Number analyzed (Participants) | 34 | 29 | 31 | 44
Participants
  Week 24 | 23 | 14 | 13 | 23
  Week 52: number analyzed (Participants) | 15 | 16 | 17 | 14
  Week 52 | 8 | 4 | 7 | 6

8. Secondary Outcome: Number of Participants With an Improvement From Baseline in Tender and Swollen Joint Count ≥ 50% at Weeks 8, 12, 24, 36, and 52 in Participants With ≥ 6 Tender and Swollen Joints in Hands and Wrists
Description: The swollen and tender join count assessments were performed at the site by an experienced independent and blinded joint evaluator.
  Joints in hands and wrists were scored for the simultaneous presence (1) or absence (0) of swelling and tenderness. Scores ranged from 0-28. A higher score indicates more severe disease.
Time Frame: Weeks 8, 12, 24, 36 and 52
Population: Full Analysis Set: Full Analysis Set: Included all participants randomized in the study. Only participants who had ≥ 6 tender and swollen joints involving hands and wrists at baseline and the opportunity to complete the visit by the date of the study termination decision being communicated to sites were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Efavaleukin Alfa Low Dose | Efavaleukin Alfa Medium Dose | Efavaleukin Alfa High Dose
Number analyzed (Participants) | 22 | 16 | 20 | 27
Participants
  Week 8 | 16 | 8 | 8 | 13
  Week 12: number analyzed (Participants) | 22 | 14 | 19 | 25
  Week 12 | 16 | 7 | 7 | 13
  Week 24: number analyzed (Participants) | 19 | 13 | 18 | 20
  Week 24 | 13 | 9 | 9 | 11
  Week 36: number analyzed (Participants) | 16 | 13 | 17 | 8
  Week 36 | 11 | 8 | 8 | 3
  Week 52: number analyzed (Participants) | 8 | 7 | 12 | 4
  Week 52 | 2 | 1 | 7 | 3

9. Secondary Outcome: Number of Participants With an Improvement From Baseline in Cutaneous Lupus Erythematosus Area and Severity Index (CLASI) Activity Score ≥ 50% at Week 8, 12, 24, 36, and 52 in Participants With a CLASI Activity Score ≥ 8 at Baseline
Description: The CLASI consists of 2 scores, the first summarizes the activity of the disease while the second is a measure of the damage done by the disease. Activity is scored based on erythema, scale/hyperkeratosis, mucous membrane involvement, acute hair loss and non-scarring alopecia. The total score ranges from 0-70, with higher scores indicating more severe disease.
Time Frame: Weeks 8, 12, 24, 36 and 52
Population: Full Analysis Set: Included all participants randomized in the study. Only participants who had a CLASI activity score ≥ 8 at baseline and the opportunity to complete the visit by the date of the study termination decision being communicated to sites were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Efavaleukin Alfa Low Dose | Efavaleukin Alfa Medium Dose | Efavaleukin Alfa High Dose
Number analyzed (Participants) | 18 | 8 | 14 | 17
Participants
  Week 8 | 2 | 1 | 5 | 9
  Week 12: number analyzed (Participants) | 18 | 8 | 12 | 17
  Week 12 | 6 | 2 | 5 | 7
  Week 24: number analyzed (Participants) | 16 | 8 | 12 | 12
  Week 24 | 4 | 4 | 5 | 6
  Week 36: number analyzed (Participants) | 11 | 8 | 10 | 8
  Week 36 | 5 | 5 | 4 | 5
  Week 52: number analyzed (Participants) | 6 | 4 | 9 | 6
  Week 52 | 3 | 0 | 3 | 3

10. Secondary Outcome: Annualized Flare Rate Over 52 Weeks
Description: A flare was defined as a BILAG score designation of "worse" or "new" resulting in a B score in ≥ 2 organs or an A score in ≥ 1 organ. The BILAG index evaluates disease activity in 9 separate organ systems. Each of the organ systems are allocated an alphabetical score of A (most active), B (moderate activity), C (minor activity), D (stable) or E (never present).
  The annualized flare rate was calculated as the number of flares divided by the flare exposure time in days multiplied by 365.25.
Time Frame: Up to 52 weeks
Population: Full Analysis Set: Included all participants randomized in the study.
Measure: Number; unit: flares per participant-year
Arm/Group | Placebo | Efavaleukin Alfa Low Dose | Efavaleukin Alfa Medium Dose | Efavaleukin Alfa High Dose
Number analyzed (Participants) | 41 | 35 | 34 | 58
flares per participant-year | 0.3 | 0.5 | 0.7 | 0.4

11. Secondary Outcome: Change From Baseline in Fatigue Standardized Score Using the Patient-Reported Outcome Measurement Information System (PROMIS) Fatigue Short Form (SF) 7a Instrument at Week 12, 24, 36 and 52
Description: The PROMIS Fatigue SF 7a assesses the experience of fatigue as well as its impact on physical, mental and social activities. The score ranges from 7 to 35, with higher scores indicating more fatigue. A negative change from baseline indicates a reduction in fatigue.
  Efficacy data collected after the study termination decision date were censored and excluded from analyses for that particular visit.
Time Frame: Baseline to Week 12, 24, 36 and 52
Population: Full Analysis Set: Included all participants randomized in the study and had observed data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Efavaleukin Alfa Low Dose | Efavaleukin Alfa Medium Dose | Efavaleukin Alfa High Dose
Number analyzed (Participants) | 37 | 27 | 24 | 46
score on a scale
  Week 12 | -4.12 (7.91) | -5.52 (5.04) | -5.78 (8.39) | -4.74 (9.60)
  Week 24: number analyzed (Participants) | 32 | 24 | 22 | 33
  Week 24 | -5.24 (8.05) | -4.95 (8.72) | -4.62 (8.03) | -7.17 (7.01)
  Week 36: number analyzed (Participants) | 23 | 21 | 14 | 19
  Week 36 | -3.20 (10.70) | -5.77 (7.09) | -5.32 (8.90) | -5.34 (10.61)
  Week 52: number analyzed (Participants) | 8 | 7 | 11 | 10
  Week 52 | -3.29 (7.64) | -8.44 (4.21) | -6.97 (14.20) | -5.47 (13.97)

12. Secondary Outcome: Change From Baseline in the Physical Component Score of the Medical Outcomes Short Form-36 Questionnaire Version 2 (SF-36V2) at Week 12, 24, 36 and 52
Description: The SF-36v2 contains 36 items and yields assessments of 8 domains of health-related quality of life:
  1. Limitations in physical activities because of health problems.
  2. Limitations in social activities because of physical or emotional problems.
  3. Limitations in usual role activities because of physical health problems.
  4. Bodily pain.
  5. General mental health (psychological distress and well-being).
  6. Limitations in usual role activities because of emotional problems.
  7. Vitality (energy and fatigue).
  8. General health perceptions.
  The scores from the 8 domains will be evaluated independently and aggregated into 2 norm-based summary component measures of physical and mental health. The recall period is the past 7 days. The score ranges from 0-100 for the summary components and for each domain, with higher scores indicating better outcomes. A positive change from baseline indicates an improvement in outcomes.
Time Frame: Baseline to Week 12, 24, 36 and 52
Population: Full Analysis Set: Included all participants randomized in the study and had observed data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Efavaleukin Alfa Low Dose | Efavaleukin Alfa Medium Dose | Efavaleukin Alfa High Dose
Number analyzed (Participants) | 37 | 27 | 24 | 46
score on a scale
  Week 12 | 4.349 (7.526) | 6.016 (7.854) | 6.450 (6.701) | 2.615 (7.622)
  Week 24: number analyzed (Participants) | 32 | 24 | 22 | 33
  Week 24 | 6.709 (7.520) | 5.544 (7.624) | 4.726 (7.058) | 5.136 (8.351)
  Week 36: number analyzed (Participants) | 23 | 21 | 14 | 19
  Week 36 | 5.391 (9.040) | 6.576 (6.331) | 7.524 (8.988) | 3.648 (8.269)
  Week 52: number analyzed (Participants) | 8 | 7 | 11 | 10
  Week 52 | 3.678 (2.958) | 6.206 (4.144) | 8.724 (9.159) | 6.252 (12.226)

13. Secondary Outcome: Change From Baseline in the Mental Component Score of the SF-36V2 at Week 12, 24, 36 and 52
Description: as for outcome 12
Time Frame: Baseline to Week 12, 24, 36 and 52
Population: Full Analysis Set: Included all participants randomized in the study and had observed data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Efavaleukin Alfa Low Dose | Efavaleukin Alfa Medium Dose | Efavaleukin Alfa High Dose
Number analyzed (Participants) | 37 | 27 | 24 | 46
score on a scale
  Week 12 | 5.079 (11.395) | 0.080 (10.789) | 3.087 (11.651) | 1.867 (9.092)
  Week 24: number analyzed (Participants) | 32 | 24 | 22 | 33
  Week 24 | 6.510 (12.498) | 0.498 (10.902) | 1.585 (9.032) | 3.959 (9.220)
  Week 36: number analyzed (Participants) | 23 | 21 | 14 | 19
  Week 36 | 5.587 (14.482) | -0.118 (10.560) | 3.129 (12.141) | 0.564 (13.586)
  Week 52: number analyzed (Participants) | 8 | 7 | 11 | 10
  Week 52 | 4.781 (8.485) | 1.106 (9.633) | -1.813 (16.608) | -2.163 (13.023)

14. Secondary Outcome: Change From Baseline in the Physical Functioning Domain Score of the SF-36V2 at Week 12, 24, 36 and 52
Description: as for outcome 12
Time Frame: Baseline to Week 12, 24, 36 and 52
Population: Full Analysis Set: Included all participants randomized in the study and had observed data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Efavaleukin Alfa Low Dose | Efavaleukin Alfa Medium Dose | Efavaleukin Alfa High Dose
Number analyzed (Participants) | 37 | 27 | 24 | 46
score on a scale
  Week 12 | 14.460 (21.532) | 7.963 (15.888) | 14.165 (22.489) | 5.761 (22.034)
  Week 24: number analyzed (Participants) | 32 | 24 | 22 | 33
  Week 24 | 20.469 (23.048) | 6.876 (20.998) | 14.545 (21.816) | 10.607 (24.036)
  Week 36: number analyzed (Participants) | 23 | 21 | 14 | 19
  Week 36 | 13.477 (26.261) | 10.713 (20.078) | 16.786 (29.910) | 9.736 (29.603)
  Week 52: number analyzed (Participants) | 8 | 7 | 11 | 10
  Week 52 | 8.750 (14.083) | 15.714 (13.973) | 18.183 (28.919) | 15.001 (31.622)

15. Secondary Outcome: Change From Baseline in the Social Role Functioning Domain Score of the SF-36V2 at Week 12, 24, 36 and 52
Description: as for outcome 12
Time Frame: Baseline to Week 12, 24, 36 and 52
Population: Full Analysis Set: Included all participants randomized in the study and had observed data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Efavaleukin Alfa Low Dose | Efavaleukin Alfa Medium Dose | Efavaleukin Alfa High Dose
Number analyzed (Participants) | 37 | 27 | 24 | 46
score on a scale
  Week 12 | 15.54 (29.82) | 9.72 (22.29) | 7.81 (26.79) | 2.17 (21.46)
  Week 24: number analyzed (Participants) | 32 | 24 | 22 | 33
  Week 24 | 21.88 (33.15) | 13.02 (23.16) | 3.98 (24.52) | 9.47 (25.39)
  Week 36: number analyzed (Participants) | 23 | 21 | 14 | 19
  Week 36 | 13.04 (38.71) | 8.93 (26.26) | 16.96 (32.75) | 1.32 (29.14)
  Week 52: number analyzed (Participants) | 8 | 7 | 11 | 10
  Week 52 | 10.94 (28.69) | 21.43 (20.04) | 5.68 (35.95) | -1.25 (36.54)

16. Secondary Outcome: Change From Baseline in the Physical Role Functioning Domain Score of the SF-36V2 at Week 12, 24, 36 and 52
Description: as for outcome 12
Time Frame: Baseline to Week 12, 24, 36 and 52
Population: Full Analysis Set: Included all participants randomized in the study and had observed data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Efavaleukin Alfa Low Dose | Efavaleukin Alfa Medium Dose | Efavaleukin Alfa High Dose
Number analyzed (Participants) | 37 | 27 | 24 | 46
score on a scale
  Week 12 | 12.838 (24.516) | 15.509 (26.081) | 13.802 (22.571) | 6.929 (21.899)
  Week 24: number analyzed (Participants) | 32 | 24 | 22 | 33
  Week 24 | 18.359 (22.221) | 14.323 (26.290) | 9.091 (20.479) | 15.909 (23.804)
  Week 36: number analyzed (Participants) | 23 | 21 | 14 | 19
  Week 36 | 11.685 (26.935) | 14.881 (26.917) | 15.179 (24.966) | 7.895 (29.377)
  Week 52: number analyzed (Participants) | 8 | 7 | 11 | 10
  Week 52 | 11.719 (15.468) | 18.750 (14.878) | 19.318 (25.381) | 6.875 (35.041)

17. Secondary Outcome: Change From Baseline in the Bodily Pain Domain Score of the SF-36V2 at Week 12, 24, 36 and 52
Description: as for outcome 12
Time Frame: Baseline to Week 12, 24, 36 and 52
Population: Full Analysis Set: Included all participants randomized in the study and had observed data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Efavaleukin Alfa Low Dose | Efavaleukin Alfa Medium Dose | Efavaleukin Alfa High Dose
Number analyzed (Participants) | 37 | 27 | 24 | 46
score on a scale
  Week 12 | 13.6 (25.1) | 13.7 (23.0) | 18.8 (22.6) | 10.2 (23.0)
  Week 24: number analyzed (Participants) | 32 | 24 | 22 | 33
  Week 24 | 20.4 (26.6) | 14.3 (21.5) | 13.8 (23.1) | 18.4 (26.6)
  Week 36: number analyzed (Participants) | 23 | 21 | 14 | 19
  Week 36 | 22.0 (26.3) | 19.5 (20.7) | 24.6 (33.0) | 15.4 (23.3)
  Week 52: number analyzed (Participants) | 8 | 7 | 11 | 10
  Week 52 | 10.4 (7.7) | 11.1 (17.1) | 17.9 (29.7) | 16.7 (37.1)

18. Secondary Outcome: Change From Baseline in the Mental Health Domain Score of the SF-36V2 at Week 12, 24, 36 and 52
Description: as for outcome 12
Time Frame: Baseline to Week 12, 24, 36 and 52
Population: Full Analysis Set: Included all participants randomized in the study and had observed data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Efavaleukin Alfa Low Dose | Efavaleukin Alfa Medium Dose | Efavaleukin Alfa High Dose
Number analyzed (Participants) | 37 | 27 | 24 | 46
score on a scale
  Week 12 | 8.2 (19.3) | 1.3 (18.7) | 9.4 (22.5) | 5.2 (17.4)
  Week 24: number analyzed (Participants) | 32 | 24 | 22 | 33
  Week 24 | 12.0 (21.2) | 3.8 (22.4) | 7.5 (19.6) | 9.4 (17.8)
  Week 36: number analyzed (Participants) | 23 | 21 | 14 | 19
  Week 36 | 9.6 (23.2) | -1.9 (18.4) | 6.4 (22.6) | 6.6 (24.3)
  Week 52: number analyzed (Participants) | 8 | 7 | 11 | 10
  Week 52 | 7.5 (16.7) | -2.1 (22.7) | 0.5 (33.0) | 1.5 (28.5)

19. Secondary Outcome: Change From Baseline in the Emotional Role Domain Score of the SF-36V2 at Week 12, 24, 36 and 52
Description: as for outcome 12
Time Frame: Baseline to Week 12, 24, 36 and 52
Population: Full Analysis Set: Included all participants randomized in the study and had observed data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Efavaleukin Alfa Low Dose | Efavaleukin Alfa Medium Dose | Efavaleukin Alfa High Dose
Number analyzed (Participants) | 37 | 27 | 24 | 46
score on a scale
  Week 12 | 13.964 (27.781) | -3.704 (23.036) | 4.514 (26.236) | 3.804 (23.812)
  Week 24: number analyzed (Participants) | 32 | 24 | 22 | 33
  Week 24 | 16.926 (29.820) | -5.208 (23.417) | 3.031 (23.223) | 8.333 (25.769)
  Week 36: number analyzed (Participants) | 23 | 21 | 14 | 19
  Week 36 | 17.028 (35.129) | 5.952 (24.029) | 6.548 (29.810) | -0.440 (33.847)
  Week 52: number analyzed (Participants) | 8 | 7 | 11 | 10
  Week 52 | 9.375 (18.057) | 8.334 (14.433) | -2.273 (33.144) | -9.168 (32.972)

20. Secondary Outcome: Change From Baseline in the Vitality Domain Score of the SF-36V2 at Week 12, 24, 36 and 52
Description: as for outcome 12
Time Frame: Baseline to Week 12, 24, 36 and 52
Population: Full Analysis Set: Included all participants randomized in the study and had observed data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Efavaleukin Alfa Low Dose | Efavaleukin Alfa Medium Dose | Efavaleukin Alfa High Dose
Number analyzed (Participants) | 37 | 27 | 24 | 46
score on a scale
  Week 12 | 10.642 (20.405) | 12.037 (21.225) | 15.365 (23.384) | 7.609 (20.536)
  Week 24: number analyzed (Participants) | 32 | 24 | 22 | 33
  Week 24 | 13.477 (23.283) | 8.333 (23.936) | 8.523 (20.912) | 12.879 (19.884)
  Week 36: number analyzed (Participants) | 23 | 21 | 14 | 19
  Week 36 | 11.685 (26.935) | 6.548 (19.811) | 14.732 (23.718) | 5.592 (22.812)
  Week 52: number analyzed (Participants) | 8 | 7 | 11 | 10
  Week 52 | 15.625 (19.480) | 4.464 (22.160) | 9.659 (28.141) | 13.750 (26.484)

21. Secondary Outcome: Change From Baseline in the General Health Domain Score of the SF-36V2 at Week 12, 24, 36 and 52
Description: as for outcome 12
Time Frame: Baseline to Week 12, 24, 36 and 52
Population: Full Analysis Set: Included all participants randomized in the study and had observed data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Efavaleukin Alfa Low Dose | Efavaleukin Alfa Medium Dose | Efavaleukin Alfa High Dose
Number analyzed (Participants) | 37 | 27 | 24 | 46
score on a scale
  Week 12 | 5.2 (15.8) | 6.1 (17.7) | 10.6 (15.9) | 2.6 (16.2)
  Week 24: number analyzed (Participants) | 32 | 24 | 22 | 33
  Week 24 | 9.2 (17.7) | 6.2 (19.0) | 3.8 (16.2) | 5.6 (15.3)
  Week 36: number analyzed (Participants) | 23 | 21 | 14 | 19
  Week 36 | 10.7 (16.1) | 5.6 (14.9) | 7.2 (17.2) | -2.1 (16.6)
  Week 52: number analyzed (Participants) | 8 | 7 | 11 | 10
  Week 52 | 7.5 (8.9) | 2.4 (5.9) | 6.7 (19.0) | 0.5 (29.5)

22. Secondary Outcome: Change From Baseline in the Physical Health Domain Score of the Lupus Quality of Life (LupusQoL) at Week 12, 24, 36 and 52
Description: The LupusQoL is a systemic lupus erythematosus (SLE)-specific health-related QoL instrument and consists of 8 domains:
  1. Physical health.
  2. Pain.
  3. Planning.
  4. Intimate relationships.
  5. Burden to others.
  6. Emotional health.
  7. Body image.
  8. Fatigue.
  The score for each domain ranges from 0-100, with higher scores indicating better outcomes. A positive change from baseline indicates an improvement in outcomes.
Time Frame: Baseline to Week 12, 24, 36 and 52
Population: Full Analysis Set: Included all participants randomized in the study and had observed data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Efavaleukin Alfa Low Dose | Efavaleukin Alfa Medium Dose | Efavaleukin Alfa High Dose
Number analyzed (Participants) | 34 | 26 | 22 | 42
score on a scale
  Week 12 | 13.7868 (20.5586) | 12.6202 (18.9259) | 13.7784 (18.3909) | 11.5327 (22.3595)
  Week 24: number analyzed (Participants) | 29 | 23 | 20 | 30
  Week 24 | 15.5172 (23.7770) | 9.5109 (25.1501) | 15.4688 (17.7205) | 13.8542 (25.3834)
  Week 36: number analyzed (Participants) | 22 | 20 | 13 | 18
  Week 36 | 11.3636 (20.6738) | 13.4375 (20.2549) | 18.7500 (24.4404) | 5.7292 (24.3304)
  Week 52: number analyzed (Participants) | 8 | 6 | 11 | 10
  Week 52 | 9.3750 (11.8114) | 20.8333 (21.1640) | 15.6250 (27.0994) | 10.6250 (29.5437)

23. Secondary Outcome: Change From Baseline in the Pain Domain Score of the LupusQoL at Week 12, 24, 36 and 52
Description: The LupusQoL is a SLE-specific health-related QoL instrument and consists of 8 domains:
  1. Physical health.
  2. Pain.
  3. Planning.
  4. Intimate relationships.
  5. Burden to others.
  6. Emotional health.
  7. Body image.
  8. Fatigue.
  The score for each domain ranges from 0-100, with higher scores indicating better outcomes. A positive change from baseline indicates an improvement in outcomes.
Time Frame: Baseline to Week 12, 24, 36 and 52
Population: Full Analysis Set: Included all participants randomized in the study and had observed data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Efavaleukin Alfa Low Dose | Efavaleukin Alfa Medium Dose | Efavaleukin Alfa High Dose
Number analyzed (Participants) | 34 | 25 | 22 | 42
score on a scale
  Week 12 | 17.892 (22.392) | 16.333 (23.873) | 17.424 (23.975) | 13.294 (24.072)
  Week 24: number analyzed (Participants) | 29 | 22 | 20 | 30
  Week 24 | 21.264 (28.311) | 14.773 (25.708) | 11.667 (23.939) | 11.944 (28.339)
  Week 36: number analyzed (Participants) | 22 | 19 | 13 | 18
  Week 36 | 12.879 (25.423) | 17.105 (21.956) | 16.667 (30.238) | 5.556 (28.296)
  Week 52: number analyzed (Participants) | 8 | 5 | 11 | 10
  Week 52 | 14.583 (18.767) | 16.667 (8.333) | 8.333 (27.639) | 11.667 (27.833)

24. Secondary Outcome: Change From Baseline in the Planning Domain Score of the LupusQoL at Week 12, 24, 36 and 52
Description: as for outcome 23
Time Frame: Baseline to Week 12, 24, 36 and 52
Population: Full Analysis Set: Included all participants randomized in the study and had observed data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Efavaleukin Alfa Low Dose | Efavaleukin Alfa Medium Dose | Efavaleukin Alfa High Dose
Number analyzed (Participants) | 34 | 25 | 22 | 42
score on a scale
  Week 12 | 9.804 (23.071) | 17.000 (23.259) | 13.636 (23.925) | 7.143 (23.825)
  Week 24: number analyzed (Participants) | 29 | 22 | 20 | 30
  Week 24 | 11.494 (29.915) | 14.015 (28.334) | 15.833 (22.926) | 14.722 (22.391)
  Week 36: number analyzed (Participants) | 22 | 19 | 13 | 18
  Week 36 | 12.500 (30.834) | 9.211 (23.553) | 13.462 (23.457) | 5.093 (29.861)
  Week 52: number analyzed (Participants) | 8 | 5 | 11 | 10
  Week 52 | 15.625 (29.693) | 15.000 (18.066) | 10.606 (25.025) | 12.500 (27.287)

25. Secondary Outcome: Change From Baseline in the Intimate Relationship Domain Score of the LupusQoL at Week 12, 24, 36 and 52
Description: as for outcome 23
Time Frame: Baseline to Week 12, 24, 36 and 52
Population: Full Analysis Set: Included all participants randomized in the study and had observed data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Efavaleukin Alfa Low Dose | Efavaleukin Alfa Medium Dose | Efavaleukin Alfa High Dose
Number analyzed (Participants) | 21 | 18 | 16 | 29
score on a scale
  Week 12: number analyzed (Participants) | 21 | 18 | 14 | 29
  Week 12 | 17.26 (27.52) | 3.47 (22.61) | 14.29 (35.65) | 11.21 (31.04)
  Week 24: number analyzed (Participants) | 15 | 16 | 16 | 19
  Week 24 | 10.83 (35.00) | 1.56 (26.57) | 19.53 (28.86) | 13.16 (29.01)
  Week 36: number analyzed (Participants) | 16 | 15 | 11 | 12
  Week 36 | 10.94 (33.81) | -1.67 (30.20) | 11.36 (30.34) | 12.50 (15.99)
  Week 52: number analyzed (Participants) | 6 | 5 | 8 | 6
  Week 52 | 6.25 (51.08) | 0.00 (8.84) | 9.38 (35.83) | 8.33 (31.29)

26. Secondary Outcome: Change From Baseline in the Burden to Others Domain Score of the LupusQoL at Week 12, 24, 36 and 52
Description: as for outcome 23
Time Frame: Baseline to Week 12, 24, 36 and 52
Population: Full Analysis Set: Included all participants randomized in the study and had observed data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Efavaleukin Alfa Low Dose | Efavaleukin Alfa Medium Dose | Efavaleukin Alfa High Dose
Number analyzed (Participants) | 34 | 25 | 22 | 42
score on a scale
  Week 12 | 10.784 (28.169) | 14.333 (17.099) | 17.803 (30.134) | 6.944 (29.673)
  Week 24: number analyzed (Participants) | 29 | 22 | 20 | 30
  Week 24 | 20.115 (31.459) | 5.682 (24.719) | 12.083 (23.798) | 12.778 (29.093)
  Week 36: number analyzed (Participants) | 22 | 19 | 13 | 18
  Week 36 | 14.773 (30.530) | 10.088 (22.149) | 21.795 (22.448) | 18.519 (26.438)
  Week 52: number analyzed (Participants) | 8 | 5 | 11 | 10
  Week 52 | 16.667 (22.713) | 38.333 (19.185) | 21.212 (23.677) | 18.333 (28.273)

27. Secondary Outcome: Change From Baseline in the Emotional Health Domain Score of the LupusQoL at Week 12, 24, 36 and 52
Description: as for outcome 23
Time Frame: Baseline to Week 12, 24, 36 and 52
Population: Full Analysis Set: Included all participants randomized in the study and had observed data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Efavaleukin Alfa Low Dose | Efavaleukin Alfa Medium Dose | Efavaleukin Alfa High Dose
Number analyzed (Participants) | 34 | 25 | 22 | 42
score on a scale
  Week 12 | 9.681 (21.729) | 10.667 (19.021) | 14.962 (28.425) | 5.258 (21.465)
  Week 24: number analyzed (Participants) | 29 | 22 | 20 | 30
  Week 24 | 13.218 (26.495) | 7.765 (19.974) | 11.458 (20.894) | 9.722 (21.283)
  Week 36: number analyzed (Participants) | 22 | 19 | 13 | 18
  Week 36 | 10.038 (25.994) | 6.798 (18.799) | 20.192 (24.641) | 3.704 (30.178)
  Week 52: number analyzed (Participants) | 8 | 5 | 11 | 10
  Week 52 | 4.167 (20.534) | 13.333 (21.123) | 15.530 (27.518) | -5.000 (25.595)

28. Secondary Outcome: Change From Baseline in the Body Image Domain Score of the LupusQoL at Week 12, 24, 36 and 52
Description: as for outcome 23
Time Frame: Baseline to Week 12, 24, 36 and 52
Population: Full Analysis Set: Included all participants randomized in the study and had observed data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Efavaleukin Alfa Low Dose | Efavaleukin Alfa Medium Dose | Efavaleukin Alfa High Dose
Number analyzed (Participants) | 34 | 25 | 22 | 42
score on a scale
  Week 12 | 9.6 (26.5) | 9.0 (18.7) | 4.1 (34.0) | 4.6 (26.6)
  Week 24: number analyzed (Participants) | 29 | 22 | 20 | 30
  Week 24 | 11.6 (30.6) | 2.3 (25.5) | 3.0 (28.2) | 5.2 (29.6)
  Week 36: number analyzed (Participants) | 22 | 19 | 13 | 18
  Week 36 | 6.1 (25.6) | 14.7 (21.4) | 18.8 (41.2) | 6.1 (28.0)
  Week 52: number analyzed (Participants) | 8 | 5 | 11 | 10
  Week 52 | 12.5 (33.3) | 17.0 (22.5) | 7.7 (37.4) | 5.5 (36.6)

29. Secondary Outcome: Change From Baseline in the Fatigue Domain Score of the LupusQoL at Week 12, 24, 36 and 52
Description: as for outcome 23
Time Frame: Baseline to Week 12, 24, 36 and 52
Population: Full Analysis Set: Included all participants randomized in the study and had observed data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Efavaleukin Alfa Low Dose | Efavaleukin Alfa Medium Dose | Efavaleukin Alfa High Dose
Number analyzed (Participants) | 34 | 25 | 22 | 42
score on a scale
  Week 12 | 8.456 (23.329) | 9.750 (15.104) | 15.909 (21.368) | 8.185 (21.273)
  Week 24: number analyzed (Participants) | 29 | 22 | 20 | 30
  Week 24 | 10.776 (24.600) | 7.670 (23.059) | 13.750 (20.135) | 13.542 (20.108)
  Week 36: number analyzed (Participants) | 22 | 19 | 13 | 18
  Week 36 | 5.966 (29.345) | 10.526 (17.561) | 12.019 (26.695) | 4.514 (23.853)
  Week 52: number analyzed (Participants) | 8 | 5 | 11 | 10
  Week 52 | 10.938 (15.580) | 25.000 (4.419) | 15.341 (26.274) | 16.250 (28.596)

30. Secondary Outcome: Number of Participants Who Experienced a Treatment-emergent Adverse Event (TEAE)
Description: A TEAE was defined as any untoward medical occurrence in a clinical study participant irrespective of a causal relationship with the study treatment and had emerged or worsened during treatment.
  A serious TEAE was defined as any untoward medical occurrence that, met at least 1 of the following criteria:
  * Resulted in death (fatal).
  * Was immediately life-threatening.
  * Required in-patient hospitalization or prolongation of existing hospitalization.
  * Resulted in persistent or significant disability/incapacity.
  * Was a congenital anomaly/birth defect.
  * Was any other medically important serious event.
  Clinically significant changes from baseline in laboratory values and vital signs were also recorded as TEAEs.
Time Frame: Day 1 to Week 56
Population: Safety Analysis Set: All randomized participants who received at least 1 dose of investigational product. After randomization, 1 participant received more than their planned medium dose of efavaleukin alfa in error, therefore the participant is also counted in the efavaleukin alfa high dose arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Efavaleukin Alfa Low Dose | Efavaleukin Alfa Medium Dose | Efavaleukin Alfa High Dose
Number analyzed (Participants) | 41 | 35 | 33 | 59
Participants
  TEAE | 29 | 29 | 33 | 55
  Serious TEAE | 4 | 3 | 4 | 3

31. Secondary Outcome: Serum Efavaleukin Alfa Concentrations by Timepoint
Description: Serum efavaleukin alfa concentrations by timepoint after multiple dose subcutaneous administration of efavaleukin alfa to participants with active systemic lupus erythematosus. Lower limit of quantification= 0.100 ng/mL.
Time Frame: Day 1: 6-24 and 48-96 hrs, Day 29, Day 43: 6-24 and 48-96 hrs, Day 85, Day 169, Day 253, Day 309, and Day 365
Population: The PK Concentration Analysis Set is defined as the subset of participants in the Safety Analysis Set who had at least 1 evaluable serum concentration (including results below the level of detection) of investigational product. PK concentration data will be analyzed according to the actual treatment received.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Efavaleukin Alfa Low Dose | Efavaleukin Alfa Medium Dose | Efavaleukin Alfa High Dose
Number analyzed (Participants) | 34 | 30 | 53
ng/mL
  Day 1: 6-24 hrs: number analyzed (Participants) | 34 | 29 | 53
  Day 1: 6-24 hrs | 5.46 (5.18) | 12.8 (12.3) | 27.4 (25.7)
  Day 1: 48-96 hrs: number analyzed (Participants) | 34 | 30 | 49
  Day 1: 48-96 hrs | 2.34 (2.52) | 5.93 (6.45) | 21.8 (30.5)
  Day 29: number analyzed (Participants) | 26 | 24 | 39
  Day 29 | 0.0201 (0.0649) | 0.0179 (0.0496) | 0.0699 (0.173)
  Day 43: 6-24 hrs: number analyzed (Participants) | 21 | 21 | 39
  Day 43: 6-24 hrs | 4.34 (5.55) | 13.9 (11.7) | 25.0 (22.6)
  Day 43: 48-96 hrs: number analyzed (Participants) | 23 | 21 | 41
  Day 43: 48-96 hrs | 2.80 (4.39) | 12.7 (17.2) | 18.1 (19.0)
  Day 85: number analyzed (Participants) | 15 | 17 | 27
  Day 85 | 0.0577 (0.223) | 0.00712 (0.0293) | 0.191 (0.316)
  Day 169: number analyzed (Participants) | 14 | 12 | 17
  Day 169 | 0.349 (1.10) | 0.0588 (0.133) | 0.140 (0.178)
  Day 253: number analyzed (Participants) | 18 | 7 | 11
  Day 253 | 0.530 (1.48) | 0.155 (0.221) | 0.458 (0.71)
  Day 309: number analyzed (Participants) | 9 | 9 | 3
  Day 309 | 0.252 (0.502) | 0.0558 (0.167) | 0.308 (0.533)
  Day 365: number analyzed (Participants) | 5 | 4 | 3
  Day 365 | 0.00 (0.00) | 0.00 (0.00) | 0.136 (0.236)

ADVERSE EVENTS:
Time Frame: All-cause mortality: From enrollment until the end of study; median (min, max) time on study was 38.23 (0.28, 62.93) weeks. Serious TEAEs and other TEAEs: Day 1 to Week 56.
Description: All-cause mortality is reported for all participants enrolled/randomized in the study. Treatment-emergent SAEs and TEAEs are reported for all participants who received at least one dose of study drug. After randomization, 1 participant received more than their planned medium dose of efavaleukin alfa in error, therefore the participant is also counted in the efavaleukin alfa high dose arm.
Arm/Group | Placebo | Efavaleukin Alfa Low Dose | Efavaleukin Alfa Medium Dose | Efavaleukin Alfa High Dose
All-Cause Mortality (participants affected / at risk) | 1/41 | 0/35 | 0/33 | 0/59
Serious Adverse Events (participants affected / at risk) | 4/41 | 3/35 | 4/33 | 3/59
Other Adverse Events (participants affected / at risk) | 18/41 | 27/35 | 33/33 | 48/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=41) | Efavaleukin Alfa Low Dose (N=35) | Efavaleukin Alfa Medium Dose (N=33) | Efavaleukin Alfa High Dose (N=59)
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0
Bartholin's abscess (Infections and infestations) | 0 | 0 | 1 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 2 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Anal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Brain stem infarction (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Stroke in evolution (Nervous system disorders) | 0 | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=41) | Efavaleukin Alfa Low Dose (N=35) | Efavaleukin Alfa Medium Dose (N=33) | Efavaleukin Alfa High Dose (N=59)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 2 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 3 | 2
Constipation (Gastrointestinal disorders) | 2 | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 4 | 2
Gastritis (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 3 | 2
Vomiting (Gastrointestinal disorders) | 1 | 0 | 2 | 3
Administration site inflammation (General disorders) | 0 | 2 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 2 | 0
Injection site discolouration (General disorders) | 0 | 0 | 3 | 1
Injection site erythema (General disorders) | 0 | 16 | 22 | 32
Injection site inflammation (General disorders) | 0 | 0 | 2 | 1
Injection site oedema (General disorders) | 0 | 1 | 0 | 3
Injection site pain (General disorders) | 1 | 4 | 10 | 10
Injection site pruritus (General disorders) | 1 | 7 | 16 | 17
Injection site rash (General disorders) | 0 | 4 | 7 | 13
Injection site reaction (General disorders) | 0 | 2 | 0 | 1
Injection site swelling (General disorders) | 0 | 6 | 6 | 9
Injection site urticaria (General disorders) | 0 | 0 | 4 | 2
Injection site warmth (General disorders) | 0 | 0 | 3 | 3
Pain (General disorders) | 1 | 0 | 0 | 3
Pyrexia (General disorders) | 1 | 1 | 2 | 6
Bronchitis (Infections and infestations) | 2 | 3 | 2 | 0
COVID-19 (Infections and infestations) | 2 | 4 | 5 | 6
Gastroenteritis (Infections and infestations) | 0 | 1 | 2 | 1
Influenza (Infections and infestations) | 0 | 0 | 1 | 3
Nasopharyngitis (Infections and infestations) | 0 | 2 | 2 | 3
Oral candidiasis (Infections and infestations) | 1 | 1 | 2 | 0
Pharyngitis (Infections and infestations) | 0 | 2 | 2 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 4 | 1 | 4
Upper respiratory tract infection bacterial (Infections and infestations) | 0 | 0 | 3 | 0
Urinary tract infection (Infections and infestations) | 3 | 1 | 5 | 5
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 2 | 4 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 4 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0 | 2 | 0
Headache (Nervous system disorders) | 4 | 4 | 5 | 5
Tension headache (Nervous system disorders) | 2 | 3 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 3 | 1 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 2 | 3 | 3

LIMITATIONS AND CAVEATS:
This study was discontinued early due to meeting predefined futility criteria at its third interim analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2023-03-06): https://cdn.clinicaltrials.gov/large-docs/37/NCT04680637/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-25): https://cdn.clinicaltrials.gov/large-docs/37/NCT04680637/SAP_001.pdf